CLINICAL TRIAL: NCT05836753
Title: Efficacy and Safety of Sarecycline in Patients With Acute Ischemic Stroke After Reperfusion Therapy: A Phase II, Randomized, Multicenter, Double-blind, Single Dose, Placebo-controlled Parallel Trial
Brief Title: Efficacy and Safety of Sarecycline in Patients With Acute Ischemic Stroke After Reperfusion Therapy
Acronym: ESPRIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2023-026-01
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Ischemic Stroke, Acute
Keywords: Ischemic Stroke, Sarecycline
MeSH Terms: conditions — Ischemic Stroke | interventions — sarecycline

STUDY DESIGN:
Intervention Model Description: This trial was a prospective, randomized, multicenter, double-blind, placebo-controlled parallel trial. Subjects were randomly assigned according to the ratio of the experimental group: control group =2:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Sarecycline drug used in the study is indistinguishable from the Sarecycline placebo (the shape, color, and appearance are identical).
  In addition, to ensure the blind method, the drug packaging and batch numbers of the two groups are identical, and the packaging batch numbers are uniformly marked.
  During the implementation of the study, except for the authorized personnel of the company's supply chain, research management department, and subject security department, members of each research execution group, research center personnel, and CRO data processing personnel cannot view the randomization scheme.
  The blind method was also used to evaluate the outcome. The subjects were randomly divided into groups and blinded to the members of the adjudication committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sarecycline treatment group (Active Comparator): The first dose should be given immediately after randomization (within 30 minutes); Take one tablet once a day for 7 days continuously (the patient with dysphagia will be administrated through a nasal feeding tube).
  Interventions: Drug: Sarecycline Tablet
- Sarecycline placebo control group (Placebo Comparator): The control group received Sarecycline placebo tablets (each containing Sarecycline 0 mg) in the same way as the experimental group.
  Interventions: Drug: Placebo tablets of Sarecycline tablets

INTERVENTIONS:
Drug: Sarecycline Tablet — Each tablet contained 100 mg of Sarecycline.
  Arms: Sarecycline treatment group
Drug: Placebo tablets of Sarecycline tablets — Each tablet contained 0 mg of Sarecycline.
  Arms: Sarecycline placebo control group

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of Sarecycline versus placebo in the treatment of microcirculation dysfunction after reperfusion therapy in patients with large vessel occlusion stroke.

DETAILED DESCRIPTION:
This study evaluated the efficacy and safety of 7-day Sarecycline versus placebo in patients with large vessel occlusion stroke who received reperfusion therapy within 24 hours of onset. In addition, we will explore the effect of Sarecycline versus placebo on indicators of venous thrombotic inflammation at different time points in patients with acute ischemic stroke with large vessel occlusion.

This trial was a prospective, randomized, multicenter, double-blind, placebo-controlled parallel trial. Patients with acute large vessel occlusion stroke who received reperfusion therapy within 24 hours of onset were randomly assigned according to the ratio of the experimental group: control group =2:1.

The trial was divided into three phases: screening/baseline period, treatment period, and follow-up period. The primary research objective is to evaluate the effect of Sarecycline in improving neurological deficits at 7 days in patients with acute large vessel occlusion stroke who received reperfusion therapy within 24 hours of onset.

ELIGIBILITY:
Inclusion criteria:

1. 18≤Age≤80 years old;
2. Acute large vessel occlusion (LVO) confirmed by imaging (CT+CTA+CTP/MRI+MRA), including the responsible vessel was located in the intracranial internal carotid artery, the T-shaped branch, the M1/M2 segment of the middle cerebral artery, or the A1/A2 segment of the anterior cerebral artery;
3. ASPECTS≥6;
4. 7≤NIHSS≤25,and Ia≤1;
5. Scheduled for reperfusion therapy within 24 hours of onset (including intravenous rt-PA or TNK-tPA thrombolysis (within 4.5 hours), mechanical thrombectomy, and bridging therapy);
6. First stroke or complete self-care before the onset of current stroke (mRS 0-1);
7. Patients or his/her legal representatives are able to understand and sign the informed consent.

Exclusion criteria:

1. History of pseudomembranous colitis or antibiotic-related colitis.
2. Allergic to tetracycline antibiotics or any component of the investigational drug.
3. Known to be resistant to other tetracyclines.
4. History of intracranial hemorrhagic diseases within the previous 3 months, including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/external hematoma, etc.
5. Intracranial tumors, vascular malformations, and other intracranial space-occupying lesions.
6. Bilateral or posterior circulation LVO.
7. Rare or unknown etiology of LVO, such as dissection and vasculitis.
8. Severe hepatic or renal insufficiency and various reasons for receiving dialysis before randomization (Severe hepatic insufficiency was defined as ALT >3 times the upper limit of normal value or AST >3 times the upper limit of normal value; Severe renal insufficiency refers to serum creatinine >3.0 mg/dl (265.2 μmol/L) or glomerular filtration rate<30 ml/min).
9. Bleeding tendency (including but not limited to): platelet count <100×109/L; Oral warfarin, INR > 2; Received heparin within previous 48 hours, APTT≥35s; Hereditary hemorrhagic diseases, such as hemophilia.
10. Received any of the following treatments within the previous 3 months: systemic retinoic acid, androgen/antiandrogen therapy (e.g., anabolic steroids, andiolactone).
11. Refractory hypertension that is difficult to control with medication (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg).
12. History of intracranial or spinal surgery within the previous 3 months; History of therapeutical surgery or major physical trauma within the previous 1 month.
13. Have other investigator-evaluated contraindications of reperfusion therapy.
14. Women of childbearing age who do not use effective contraception and have no negative pregnancy test records; Women during lactation and pregnancy.
15. Life expectancy of fewer than 6 months due to advanced stage of any comorbidity.
16. Participated in other interventional clinical trials within the previous 3 months.
17. Other conditions that are not suitable for participating in this clinical trial, such as inability to understand and/or follow the research procedures due to mental, cognitive, emotional, or physical disorders, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-07 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes of NIHSS score between baseline and at 7 days after randomization. | at 7 days after randomization
  National Institute of Health stroke scale (NIHSS 0-42 scores; higher scores mean a worse outcome）

SECONDARY OUTCOMES:
Changes of NIHSS score between baseline and within 2 hours after reperfusion. | within 2 hours after reperfusion
  National Institute of Health stroke scale (NIHSS 0-42 scores; higher scores mean a worse outcome）al Institute of Health stroke scale (NIHSS 0-42 scores; higher scores mean a worse outcome） National Institute of Health stroke scale (NIHSS 0-42 scores; higher scores mean a worse outcome）
Changes of NIHSS score between baseline and 72 hours after randomization. | at 72 hours after randomization
  National Institute of Health stroke scale (NIHSS 0-42 scores; higher scores mean a worse outcome）
Early neurological deterioration at 72 hours after randomization. | at 72 hours after randomization.
  Early neurological deterioration
Early neurological deterioration at 7 days after randomization. | at 7 days after randomization
  Early neurological deterioration
Changes of infarction volume between baseline and at 72 hours after randomization. | at 72 hours after randomization
  Infarction volume
Changes of cerebral blood perfusion between baseline and at 72 hours after randomization. | at 72 hours after randomization
  Cerebral blood perfusion evaluated by CTP
Changes of collateral circulation compensation between baseline and at 72 hours after randomization. | at 72 hours after randomization
  Collateral circulation compensation
Modified Rankin Scale (mRS) score at 90 days after randomization. | at 90 days after randomization
  Modified Rankin Scale (mRS 0-5 scores; higher scores mean a worse outcome）
Quality of life (EQ-5D) score at 90 days after randomization. | at 90 days after randomization
  EuroQol Five Dimensions Questionnaire
The proportion of combined vascular events (recurrent stroke, myocardial infarction, and vasogenic death) at 90 days after randomization. | at 90 days after randomization
  Combined vascular events (recurrent stroke, myocardial infarction, and vasogenic death)

OTHER OUTCOMES:
Venous thrombotic inflammation indicators compare with baseline. | within 2 hours after reperfusion therapy.
  plasma sGPVI, sADAMTS 13, sCD40L levels.
Venous thrombotic inflammation indicators compare with baseline. | at 24±2 hours after randomization.
  plasma sGPVI, sADAMTS 13, sCD40L levels.
Venous thrombotic inflammation indicators compare with baseline. | at 10±1 days after randomization
  plasma sGPVI, sADAMTS 13, sCD40L levels.
Symptomatic intracranial hemorrhage. | at 24±2 hours after randomization
  Heidelberg hemorrhage classification.
Symptomatic intracranial hemorrhage. | at 10±1 day after randomization
  Heidelberg hemorrhage classification.
Any bleeding event. | at 90±7 days after randomization.
  Any bleeding event was defined as any hemorrhagic event that occurred in the opinion of the investigator, including subcutaneous bleeding, gingival bleeding, gastrointestinal bleeding, intracranial bleeding, and other hemorrhagic events.
Vascular death. | At 90±7 days after randomization.
  Vascular origin including death due to stroke death, sudden cardiac death, death due to acute myocardial infarction and death due to heart failure, pulmonary embolism, heart/cerebrovascular intervention operation (has nothing to do with acute MI) or surgery death and death from cardiovascular causes other(such as: sudden cardiac death had nothing to do with arrhythmia, aneurysm rupture, or peripheral artery disease).
Overall mortality. | At 90±7 days after randomization.
  Death caused by any circumstances.
Investigator-reported adverse events/serious adverse events. | At 90±7 days of randomization.
  Absolute platelet value ≤100×10^9/L, high sensitivity reaction and kidney failure.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, PhD，MD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, , China
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

REFERENCES:
- [Result] Smith WS, Lev MH, English JD, Camargo EC, Chou M, Johnston SC, Gonzalez G, Schaefer PW, Dillon WP, Koroshetz WJ, Furie KL. Significance of large vessel intracranial occlusion causing acute ischemic stroke and TIA. Stroke. 2009 Dec;40(12):3834-40. doi: 10.1161/STROKEAHA.109.561787. Epub 2009 Oct 15. PMID 19834014
- [Result] Hussein HM, Georgiadis AL, Vazquez G, Miley JT, Memon MZ, Mohammad YM, Christoforidis GA, Tariq N, Qureshi AI. Occurrence and predictors of futile recanalization following endovascular treatment among patients with acute ischemic stroke: a multicenter study. AJNR Am J Neuroradiol. 2010 Mar;31(3):454-8. doi: 10.3174/ajnr.A2006. Epub 2010 Jan 14. PMID 20075087
- [Result] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Result] van Horn N, Kniep H, Leischner H, McDonough R, Deb-Chatterji M, Broocks G, Thomalla G, Brekenfeld C, Fiehler J, Hanning U, Flottmann F. Predictors of poor clinical outcome despite complete reperfusion in acute ischemic stroke patients. J Neurointerv Surg. 2021 Jan;13(1):14-18. doi: 10.1136/neurintsurg-2020-015889. Epub 2020 May 15. PMID 32414889
- [Result] Casetta I, Fainardi E, Saia V, Pracucci G, Padroni M, Renieri L, Nencini P, Inzitari D, Morosetti D, Sallustio F, Vallone S, Bigliardi G, Zini A, Longo M, Francalanza I, Bracco S, Vallone IM, Tassi R, Bergui M, Naldi A, Saletti A, De Vito A, Gasparotti R, Magoni M, Castellan L, Serrati C, Menozzi R, Scoditti U, Causin F, Pieroni A, Puglielli E, Casalena A, Sanna A, Ruggiero M, Cordici F, Di Maggio L, Duc E, Cosottini M, Giannini N, Sanfilippo G, Zappoli F, Cavallini A, Cavasin N, Critelli A, Ciceri E, Plebani M, Cappellari M, Chiumarulo L, Petruzzellis M, Terrana A, Cariddi LP, Burdi N, Tinelli A, Auteri W, Silvagni U, Biraschi F, Nicolini E, Padolecchia R, Tassinari T, Filauri P, Sacco S, Pavia M, Invernizzi P, Nuzzi NP, Marcheselli S, Amista P, Russo M, Gallesio I, Craparo G, Mannino M, Mangiafico S, Toni D; Italian Registry of Endovascular Treatment in Acute Stroke. Endovascular Thrombectomy for Acute Ischemic Stroke Beyond 6 Hours From Onset: A Real-World Experience. Stroke. 2020 Jul;51(7):2051-2057. doi: 10.1161/STROKEAHA.119.027974. Epub 2020 Jun 17. PMID 32568647
- [Result] Ng FC, Coulton B, Chambers B, Thijs V. Persistently Elevated Microvascular Resistance Postrecanalization. Stroke. 2018 Oct;49(10):2512-2515. doi: 10.1161/STROKEAHA.118.021631. PMID 30355104
- [Result] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Result] McGarry T, Biniecka M, Veale DJ, Fearon U. Hypoxia, oxidative stress and inflammation. Free Radic Biol Med. 2018 Sep;125:15-24. doi: 10.1016/j.freeradbiomed.2018.03.042. Epub 2018 Mar 27. PMID 29601945
- [Result] Stoll G, Nieswandt B. Thrombo-inflammation in acute ischaemic stroke - implications for treatment. Nat Rev Neurol. 2019 Aug;15(8):473-481. doi: 10.1038/s41582-019-0221-1. Epub 2019 Jul 1. PMID 31263257
- [Result] Kollikowski AM, Schuhmann MK, Nieswandt B, Mullges W, Stoll G, Pham M. Local Leukocyte Invasion during Hyperacute Human Ischemic Stroke. Ann Neurol. 2020 Mar;87(3):466-479. doi: 10.1002/ana.25665. Epub 2020 Jan 16. PMID 31899551
- [Result] El Amki M, Wegener S. Improving Cerebral Blood Flow after Arterial Recanalization: A Novel Therapeutic Strategy in Stroke. Int J Mol Sci. 2017 Dec 9;18(12):2669. doi: 10.3390/ijms18122669. PMID 29232823
- [Result] Bustamante A, Ning M, Garcia-Berrocoso T, Penalba A, Boada C, Simats A, Pagola J, Ribo M, Molina C, Lo E, Montaner J. Usefulness of ADAMTS13 to predict response to recanalization therapies in acute ischemic stroke. Neurology. 2018 Mar 20;90(12):e995-e1004. doi: 10.1212/WNL.0000000000005162. Epub 2018 Feb 14. PMID 29444972
- [Result] Shi K, Tian DC, Li ZG, Ducruet AF, Lawton MT, Shi FD. Global brain inflammation in stroke. Lancet Neurol. 2019 Nov;18(11):1058-1066. doi: 10.1016/S1474-4422(19)30078-X. Epub 2019 Jul 8. PMID 31296369